CLINICAL TRIAL: NCT03281109
Title: The Effect of Menstrual Cycle on Periodontium
Brief Title: The Effect of Menstrual Cycle On IL-6, TNF-α And Periodontal Status
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacer Sahin Aydinyurt, assistant professor, Yuzuncu Yil University
Other Study IDs: YuzuncuYıl4
Record Dates: First submitted 2017-08-16; First posted 2017-09-13 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Menstrual Cycle-Associated Gingivitis
Keywords: menstrual cycle; gingivitis; interleukin 1; tumor necrosis factor alpha
MeSH Terms: conditions — Gingivitis | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnosis — diagnosis with ELISA

SUMMARY:
Aim: Women's menstrual cycle is controlled by the secretion of sex hormones. Sex steroid hormones are thought to be affect to periodontal tissues, wound healing, periodontal disease progression and bone turn over. The aim the study is to evaluate clinical periodontal parameters and interleukin- 6 (IL-6) and tumor necrosis factor alpha (TNF-α) levels in gingival crevicular fluid (GCF) in menstrual cycle.

Material and methods: Twenty-five patients were included in this study clinical periodontal parameters and levels of IL-6 and TNF α in gingival crevicular fluid were evaluated at three periods of menstrual cycle (menstruation day (MD)-ovulation day(OD)-premenstruation day (PmD)). Levels of IL-6 and TNF α in gingival crevicular fluid were determined by ELISA.

DETAILED DESCRIPTION:
Study Population

Sixty women were initially included in this longitudinal, prospective study in Yuzuncu Yil University, Faculty of Dentistry, Department of Periodontology.

The procedure was accepted and informed consent was signed by all participants. The material and method used in the trial were accepted by the Yuzuncu Yil University Ethics Committee and were found to conform to the guidelines issued in the Declaration of Helsinki. To standardize the effect of plaque accumulation on the tested parameters, subjects were given oral hygiene instructions before the study.

Clinical Procedures, and Measurements

All subjects were scheduled for periodontal measurements and GCF sampling on the specific days determined as follows: 1) menstruation day (MD); on days 2-3 of menstruation 2) ovulation day (OD); detected by saliva fertility microscope 12-14 days of menstrual cycle and 3) premenstruation day (PmD); 22-24 days of menstruation cycle.

The subjects evaluated the study criteria in terms of the duration of a regular menstrual cycle (28 ± 3 d) and were followed up for three menstrual cycles. Five participants were excluded from the study if their menstrual cycles were longer or shorter than 28 ± 3 d for the last 12 months.

Donna ® Saliva Fertility Tester was used to detect the ovulation day. Patients also made their own fever measurement and confirmed the ovulation day. A small amount of saliva was placed onto microscope and after 5 minutes results were evaluated according to manufacturer's instructions. The outside of microscope lens cleaned with alcohol and a cotton swab after each use.

Periodontal measurements were performed for all patients at each of the three time points from index teeth. Periodontal measurements were: 1) plaque index (PI) (according to Silness and Löe index) 9: measured at six sites around each tooth; the highest score per tooth was recorded; 2) gingival index (GI) (according to Löe and Silness index) 10: measured at six sites around each tooth; the highest score per tooth was recorded; 3) probing depth (PD): measured at six sites around each tooth.

The GCF samples were obtained for 30 seconds from the mesiobuccal gingival sulcus of teeth using periodontal paper strips . The samples were taken 3 hours after the patients brush their teeth in the morning.

To avoid irritation of the periodontal pocket epithelium, the clinical measurements were obtained after the GCF samples collecting. The area was isolated with cotton rolls. All paper strips were stored in phosphate buffered solution. Paper points contaminated with blood and saliva were not used for study. GCF samples were stored at -80 °C for laboratory analyses. GCF samples were analyzed for IL-6 and TNF-α using commercially available sandwich enzyme-linked immunosorbent assay according to the manufacturer's instructions. Results were reported as concentrations of IL-6 and TNF-α in GCF.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria were:

1. premenopausal women, age 20-35 to years;
2. normal and steady menstrual cycle (25 to 31 days long);
3. available for clinical examination;
4. non-smoking;
5. antibiotic therapy or use of nonsteroidal anti-inflammatory drugs within the past 6 months;
6. healthy systemic status;
7. normal body mass index;
8. healthy periodontium.

Exclusion Criteria: Exclusion criteria were as follows:

1. pregnancy;
2. use of oral contraceptives;
3. metabolic or systemic condition that might affect the periodontium;
4. antibiotic therapy or use of nonsteroidal anti-inflammatory drugs within the past 6 months;
5. periodontitis;
6. smoking and
7. with the diagnosis of polycystic over or hyperandrogenism according to Rotterdam diagnostic criteria

Ages: 20 Years to 29 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only Female
Study Population: 25 women were included in this longitudinal, prospective study in Yuzuncu Yil University, Faculty of Dentistry, Department of Periodontology
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
periodontal clinical parameters | 1 menstrual cycle (approximately 1 month) every patient follow up
  gingival index: according to Silness and Löe gingival index plaque index: according to Löe and Silness plaque index probing depth the distance between gingival margin to periodontal sulcus bottom (mm) IL-6 concentration (pg/microliter) TNF- alpha concentration (pg/microliter)

CONTACTS AND LOCATIONS:
Overall Officials: hacer sahin aydinyurt, Study Director — yuzuncu yil universtiy
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided